CLINICAL TRIAL: NCT04080843
Title: An Open, Single Arm, Multicenter, Exploratory Phase II Clinical Trial of Anlotinib Hydrochloride Capsules Combined With CAPEOX in RAS and BRAF Wild-type Patients With Metastatic Colorectal Carcinoma as 1st Therapy
Brief Title: Anlotinib Hydrochloride Capsules Combined With CAPEOX in RAS and BRAF Wild-type mCRC Patients
Acronym: ALTER-C-002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ding Ke-Feng, Clinical professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-C-002
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Cancer; RAS and BRAF Wild-type; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): Patients in the study group will receive the following treatment:
  21 days as a treatment cycle, Anlotinib 12 mg/day, Orally(D1-D14); Capecitabine 850 mg/m2,Orally(D1-D14), Bid; Oxaliplatin 130 mg/m2, iv(D1).
  If anlotinib is not tolerated(except Hand-foot skin reaction), the dose can be reduced to 10mg or 8mg ,until un-tolerable toxicity again. After 6 cycles of combined therapy, patients will receive capecitabine and anlotinib as maintenance therapy until tumor progression.
  Interventions: Drug: Anlotinib Hydrochloride; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib Hydrochloride is a capsule in the form of 8 mg ,10 mg and 12 mg, orally, once daily, 2 weeks on/1 week off.
Drug: Capecitabine — Capecitabine is a capsule in the form of 500 mg, orally, 850 mg/m2, twice daily, 2 weeks on/1 week off.
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2,D1

SUMMARY:
This is an Open, Single Arm, Exploratory and Phase II Clinical Trial of Anlotinib Hydrochloride Capsules Combined With CAPEOX in RAS and BRAF wild-type patients with Metastatic Colorectal Carcinoma(CRC) as 1st Therapy. After 6 cycles of combined therapy, patients will receive capecitabine and anlotinib as maintenance therapy until tumor progression.In order to observe and evaluate the efficacy and safety of Anlotinib Hydrochloride Capsules combined with CAPEOX in treatment of patients with mCRC. The patients who are pathologically confirmed as RAS and BRAF wild-type mCRC will be enrolled.

Condition or disease Invention/treatment Phase Colorectal Cancer Drug: Anlotinib Hydrochloride Drug: Capecitabine Drug: Oxaliplatin Phase 2

DETAILED DESCRIPTION:
This is an Open, Single Arm, Exploratory and Phase II Clinical Trial of Anlotinib Hydrochloride Capsules Combined With CAPEOX in RAS and BRAF wild-type patients with Metastatic Colorectal Carcinoma(CRC) as 1st Therapy. After 6 cycles of combined therapy, patients will receive capecitabine and anlotinib as maintenance therapy until tumor progression.In order to observe and evaluate the efficacy and safety of Anlotinib Hydrochloride Capsules combined with CAPEOX in treatment of patients with Metastatic Colorectal Carcinoma(mCRC).Primary Efficacy Endpoint: Objective Response Rate (ORR), Secondary Efficacy Endpoints: Progression free survival (PFS) (According to RECIST Version 1.1), Disease Control Rate (DCR) and duration of response(DoR). Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 4.0.

ELIGIBILITY:
Inclusion Criteria:

* At least one measurable lesion (the length of spiral CT scan (> 10mm) meets the requirements of RESCIST 1.1) is found in patients with HCC confirmed by histopathology or cytology or who meet the clinical diagnostic criteria.
* ≥ 18 and ≤ 75 years of age
* ECOG performance status of 0-1
* No prior treatment for advanced disease (adjuvant therapy allowed)
* Life expectancy of at least 3 months
* The main organs are functioning normally.
* Neutrophils count =/> 1.5 x 109/L, platelets count =/> 100 x 109/L, HGB =/> 90 g/L
* total bilirubin =/< 1.5 x UNL • SGOT and SGPT =/< 2.5 x UNL (=/< 5 x UNL in patients with liver metastases)
* Creatinine =/< 1.5 x UNL
* Patients who are molecularly diagnosed as having RAS and BRAF wild-type mCRC are Histologically/cytologically confirmed as advanced, colorectal cancer.
* Subjects volunteered to join the study, signed informed consent, good compliance, with follow-up.

Exclusion Criteria:

* Pregnant or lactating women.
* Active or untreated CNS metastases as determined by CT or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments.
* Patients with hypertension who could not be well controlled by antihypertensive drugs (systolic blood pressure > 150 mmHg, diastolic blood pressure > 100 mmHg), patients with myocardial infarction, arrhythmias with poor control (including QTC interval > 450 ms) and cardiac insufficiency of grade II according to NYHA standard.
* with bleeding tendency or undergoing thrombolysis or anticoagulation therapy.
* serious uncontrolled intercurrence infection.
* Proteinuria ≥ 2+ (1.0g/24hr).
* Have evidence or a history of bleeding tendency within two months of the enrollment, regardless of seriousness.
* Within 6 months before the first treatment occurs artery/venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack) etc.
* Have a history of mental illness or psychotropic drug abuse.
* Patients with a history of immunodeficiency(or autoimmue disease), or other acquired congenital immunodeficiency diseases, or a history of organ transplantation and hematopoietic stem cell transplantation.
* Patients who are allergic to components of Capecitabine preparations, Oxaliplatin injection and anlotinib preparations.
* According to the researchers' judgment, there are serious concomitant diseases that endanger patient safety or prevent patients from completing the study.
* Patients who have received prior systemic chemotherapy, targeted therapy, immunity therapy or any medication within 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate(ORR) | Every 2 weeks until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  using RECIST version 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | every 2 weeks until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  using RECIST version 1.1
Disease control rate (DCR) | every 2 weeks until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  using RECIST version 1.1
Duration of Response (DoR) | every 2 weeks until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  using RECIST version 1.1
Safety: NCI CTC AE Version 4.0.3 | from day 1 of first dosing to 30 days after permanent discontinuation of Anlotinib
  Safety will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 4.0.3

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Xiao Q, He J, Hu H, Du J, Zhu Y, Chen J, Liu Z, Wang J, Sun L, Xu D, Li J, Liao X, Wang J, Cai Y, Cai C, Jin Z, Wang L, Yuan Y, Ding K. Phase II study of anlotinib in combination with oxaliplatin and capecitabine for patients with RAS/BRAF wild-type metastatic colorectal adenocarcinoma as the first-line therapy. BMC Med. 2022 May 6;20(1):155. doi: 10.1186/s12916-022-02357-6. PMID 35513832